CLINICAL TRIAL: NCT00672451
Title: Rhubarb and Angiotensin Converting Enzyme Inhibitor
Acronym: RACE II
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: unable to meet recruitment goal
Sponsor: Wake Forest University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00000616; 1R21AT002367-01A2 (NIH)
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Results first posted 2018-11-15 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-11

CONDITIONS: Diabetic Kidney Disease
Keywords: diabetic kidney disease; albuminuria
MeSH Terms: conditions — Diabetic Nephropathies; Albuminuria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- rhubarb extract (Experimental): will receive rhubarb extract
  Interventions: Dietary Supplement: rhubarb extract
- placebo (Placebo Comparator): receive placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: rhubarb extract — titrate rhubarb extract titrated up to 6grams daily by mouth
  Arms: rhubarb extract
Dietary Supplement: placebo — placebo titrated up to 6 pills daily as patient tolerates
  Arms: placebo

SUMMARY:
Rhubarb extract is a chinese herbal preparation that is used in china and other asian countries to treat constipation and chronic kidney disease. Use of angiotensin converting enzyme inhibitors (ACEI) in diabetic kidney disease has been shown to be beneficial in slowing progression. The purpose of this study is to determine the combined effect of rhubarb plus enalapril (an ACEI)in slowing the rate of decline of CKD in people with kidney disease from diabetes.

DETAILED DESCRIPTION:
Use of angiotensin converting enzyme inhibitors (ACEI) in diabetic nephropathy has been shown to be beneficial in slowing progression of disease. This would include use of ACEI, aggressive blood pressure and blood sugar control as well as other possible interventions. Experimental studies in chronic kidney disease (CKD) patients in China has suggested that rhubarb extract when used alone is equivalent to the protection afforded by ACEI. Furthermore when used in combination with ACEI, the renoprotective effect of rhubarb appears to be additive.

Rhubarb extract is a chinese herbal preparation that is used extensively in china and other asian countries to treat constipation and CKD. Its mechanism of action in preventing progression of CKD is uncertain but perhaps related to TGF beta and TNF alpha inhibition.

The specific aim is to determine the combined effect of rhubarb plus enalapril slowing the rate of decline of CKD (using Iothalamate GFRs) in patients in diabetes. A secondary aim would be to measure serum TGF beta concentrations over time and see if any observed decrease in the rate of decline of CKD is related to changes in TGF beta levels.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients >18 years
2. Patients with diabetic nephropathy (history of type 1 or type 2 diabetes for > 7 years, no other cause for proteinuria listed in their medical chart). This is the definition used in most peer-reviewed trials44,45 of diabetic nephropathy. We do recognize that their proteinuria could be due to some other concomitant kidney disease but the only way to confirm that is to do a kidney biopsy which is not clinically justified.
3. Proteinuria ≥ 0.5 g/day
4. Ability to sign consent form

Exclusion Criteria:

1. Pre study GFR (see section 10.7) < 20 ml/min
2. Renal disease of etiologies other than diabetes
3. Uncontrolled hypertension (Systolic BP >180 mmHg and Diastolic BP >110mm Hg)
4. Patients with history of kidney stones in past 10 years
5. Patients with active chronic liver disease (Liver enzymes ALT, AST >2.5 times normal)
6. Patients with primary small bowel disease with malabsorption, blind loop syndrome, or jejunoileal bypass surgery (may cause unabsorbed fatty acids to combine with calcium which in turn causes too much absorption of oxalate)
7. Patients with current alcohol, illicit drug use or any other condition (eg. Psychiatry disorder) that in the opinion of the investigator may interfere with the patient's ability to comply with the study
8. Pregnant women or women of child bearing potential who are unwilling to use an adequate form of contraceptive during the course of the study (ACEI may be fetotoxic)
9. Patients with significant unstable cardiovascular disease (NYHA class III and IV)
10. Patients with active malignancy
11. Uncontrolled infections.
12. Patients with a known sensitivity to the study medications (including enalapril)
13. Patients on angiotensin II receptor blockers (ARBs)
14. Microscopic or macroscopic hematuria (to rule out kidney disease other than diabetic nephropathy)
15. Patients on any herbal supplements unwilling to discontinue them
16. Severe malnutrition (serum albumin <2.6mg/dL)
17. Hyperkalemia at baseline, defined as serum potassium ≥ 5.5 mg/dL
18. Iodine allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Burkart, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Heath Sciences, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 Participants were not included in the study analysis or assigned to a group prior to termination.
Period: Overall Study
Arm/Group | Rhubarb Extract | Placebo
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rhubarb Extract | Placebo | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Albumin Concentration in Urine
Time Frame: up to 15 months
Population: Data not collected in all participants of the placebo group.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Rhubarb Extract | Placebo
Number analyzed (Participants) | 1 | 1
mg/dL | .3 (0) | 7.9 (0)

2. Secondary Outcome: Rate of Decline of GFR
Time Frame: 2 years
Population: No data collected
Arm/Group | Rhubarb Extract | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 2 years
Arm/Group | Rhubarb Extract | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

LIMITATIONS AND CAVEATS:
This study was terminated for lack of accrual. The rate of decline of GFR was not calculated as the values needed were not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes